CLINICAL TRIAL: NCT02027805
Title: A Phase I/II Multicentric Study to Determine the Safety and Efficacy of a Combination of Anti-CD3 & Anti-CD7 Ricin A Immunotoxins (T-Guard) for the Treatment of Steroid-resistant Acute Graft-versus-Host Disease.
Brief Title: Safety and Efficacy Study of T-Guard to Treat Steroid-resistant Acute GVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xenikos (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XEN/TG-001; 2013-000068-27 (EudraCT Number)
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Graft vs Host Disease
Keywords: Steroid-resistant; Graft vs Host Disease; Refractory acute Graft vs Host Disease; Hematopoietic Stem Cell Transplantation; Stem Cell Transplantation; Allogeneic Stem Cell Transplantation; Immune System Diseases; Antibodies, monoclonal; Immunotoxins; Immunosuppressive agents
MeSH Terms: conditions — Graft vs Host Disease; Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-Guard (Experimental): Four doses of T-Guard (4 mg/m2), administered at 48-hour intervals as 4 hour infusions.
  Interventions: Biological: T-Guard

INTERVENTIONS:
Biological: T-Guard
  Other Names: Combination of SPV-T3a-RTA and WT1-RTA (equal parts, w/w)

SUMMARY:
In this study, a combination of two antibodies both conjugated to a cell-killing toxin (so-called immunotoxins) will be evaluated. The antibodies are directed against T-cell antigens 'cluster of differentiation 3 antigen' (CD3) and CD7. Previous in vitro studies have demonstrated that this particular immunotoxin-combination, named T-Guard, acts synergistically in eliminating T cells with a preference for killing activated T-cells. In a subsequent clinical pilot-study, T-Guard has generated encouraging results when applied as third-line therapy for patients suffering form steroid-resistant acute Graft-versus-Host Disease (GVHD). Extensive biological and clinical responses could be noted in the absence of severe acute toxicities. Building on these results, the current study aims at evaluating the safety and efficacy of T-Guard for treating steroid-resistant GVHD when administered in an earlier phase of the disease process, i.e. as second-line instead of as third-line therapy.

DETAILED DESCRIPTION:
The experimental design is a bicentric non-controlled fixed-dose Phase I/II study. A total of 20 adult patients with acute steroid-resistant GVHD will be enrolled in a 12 months period. The treatment consists of a standard dose of 4 infusions T-Guard (4 mg/m2), given 48-hours apart over a 4-hour period. The intended follow-up period is 6 months.

The primary objective is to determine the efficacy of T-Guard, 4 weeks after the first infusion (Day 28), in inducing an objective clinical response in patients with acute GVHD refractory to standard first line corticosteroid therapy.

Secondary objectives are:

* To evaluate the overall safety and efficacy of T-Guard during the first 6 months after imitation of therapy;
* To determine the pharmacokinetic profile of T-Guard;
* To determine the immunogenicity of T-Guard.

Exploratory objectives are:

* To study the specificity and kinetics of the treatment-induced depletion and subsequent repopulation of lymphocyte subsets;
* To evaluate diagnostic and predictive GVHD biomarkers relative to treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from acute GVHD which is staged Grade II-IV according to the modified Glucksberg Criteria and progressing after 3 days, or not improving after 7 days, of methylprednisolone at a dose of 2 mg/kg per day.
* Age ≥18 years.
* Patients or an impartial witness (in case the patient is capable to provide verbal consent but not capable to sign the informed consent) should have given written informed consent.

Exclusion Criteria:

* Patients receiving concomitant investigational therapeutics for acute GVHD, including investigational agents used for GVHD prophylaxis, at the time of enrollment.
* Patients with signs or symptoms suggestive of chronic GVHD.
* Patients requiring mechanical ventilation, requiring vasopressor support, requiring hemodialysis, having serum creatinine > 266 µmol/l (> 3 mg/dl), or having a serum albumin level of 15 g/l or less.
* Patients having uncontrolled bacterial, viral or fungal infections, at the discretion of the investigator, at the start of therapy.
* Patients with current signs or symptoms of active intrapulmonary disease.
* Patients with known hypersensitivity to any of the components of the study drug.
* Female patients who are pregnant, breast feeding, or, if sexually active, unwilling to use effective birth control for the duration of the study.
* Male patients who are, if sexually active, unwilling to use effective birth control for 30 days after the last infusion.
* Patients participating in a clinical trial with another investigational product within 30 days prior to providing informed consent.
* Patients whose decision to participate might be unduly influenced by perceived expectation of gain or harm by participation, such as patients in detention due to official or legal order.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03-05 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-11-03 (Actual)

PRIMARY OUTCOMES:
Acute GVHD response rate | Day 28
  The acute GVHD response rate at 4 weeks after the first injection of T-Guard (Day 28), being defined as as the fraction of patients showing a complete or partial response (CR or PR)

SECONDARY OUTCOMES:
Safety and tolerability of T-Guard | During 6 months after initiation of treatment
  The safety and tolerability of T-Guard as assessed by evaluating Dose Limiting Toxicities (DLT's), adverse and serious adverse events reported during 6 months after initiation of treatment.
Very good partial response rate | Day 28
  The proportion of patients achieving a very good partial response rate (VGPR) of their acute GVHD at 4 weeks after the first infusion (Day 28).
Acute GVHD relapse rate | During 6 months after initiation of therapy
Incidence of chronic GVHD | During 6 months after initiation of therapy
Overall survival and progression free survival | During 6 months after initiation of treatment
Pharmacokinetic profile of T-Guard | Up to Day 9
  * Areas under the time-concentration curves (AUC);
  * Peak concentration (Cmax);
  * Time to peak concentration (Tmax);
  * Terminal-phase elimination half-life (t1/2);
  * Apparent Clearance (CL/F);
  * Steady-state volume of distribution (Vss/F).
Anti-drug-antibodies | Pre-treatment, Day 14, Day 28, Day 90, and Day 180
  The occurrence and extent of humoral responses against T-Guard (anti-drug-antibodies, ADA).
The occurrence of treatment-induced cytokine release | Day 1, 3, 5, and 7
  The occurrence of treatment-induced cytokine release, as determined by measurement of interleukin-2 (IL-2), IL-4, IL-5, IL-6, IL-8, IL-10, tumor necrosis factor-alpha (TNF-a), and interferon-gamma (IFN-g) serum levels at t = 0 (pre-dose), 1 and 4 hours after starting of each infusion.

OTHER OUTCOMES:
Kinetics and specificity of treatment-induced T cell and natural killer cell (NK cell) depletion | Up to Day 28
  Determined by the flow cytometric assessment of the number of T-, B- and NK-cells during the first 4 weeks after initiation of treatment
Composition and evolution of T-, B- and NK-cell compartments | Pre-treatment, Day 28, Day 90, and Day 180
  The flow cytometric phenotyping of lymphocyte subsets for determine the composition and evolution of the T-, B-, and NK-cells compartments at pretreatment and at 4 weeks, 3 and 6 months after the first infusion.
Composition and evolution of T-cell receptor (TCR) Vbeta repertoire | Pre-treatment, Day 28, Day 90, and Day 180
The identification and evolution of host-reactive T-cell clones | Pre-treatment, Day 28, Day 90, and Day 180
GVHD Biomarkers | Pre-treatment, Day 14, Day 28, Day 90, and Day 180
  Measurement of diagnostic and predictive GVHD biomarkers relative to treatment outcomes, including citrulline, C reactive protein (CRP), elafin, IL-8, tumor necrosis factor receptor 1 (TNFR1), interleukin 2 receptor-alpha (IL-2Ralpha), hepatocyte growth factor (HGF), and Reg3alpha.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Van der Velden, MD, PhD, Principal Investigator — Radboudumc, Nijmegen (Netherlands); Matthias Stelljes, MD, PhD, Principal Investigator — Unversity Hospital Münster, Münster (Germany)
Locations (2):
- University Hospital Münster, Münster, North Rhine-Westphalia, Germany
- Radboudumc, Nijmegen, Gelderland, Netherlands